CLINICAL TRIAL: NCT05470907
Title: South-Eastern Europe Registry for Hemoperfusion of Covid-19 ICU Patients
Brief Title: Registry for Hemoperfusion of Covid-19 ICU Patients
Acronym: HERICC
Status: Completed | Type: Observational
Sponsor: Croatian Society for Organ Support (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Vedran Premuzic, Principal Investigator, Croatian Society for Organ Support
Other Study IDs: HERICC-1982
Record Dates: First submitted 2022-07-21; First posted 2022-07-22 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Viral Disease; Critical Illness; Multi Organ Failure; Systemic Inflammatory Response Syndrome; AKI - Acute Kidney Injury
Keywords: COVID-19 Acute Respiratory Distress Syndrome; Viral Disease; Critical Illness; Multi Organ Failure; Systemic Inflammatory Response Syndrome; AKI - Acute Kidney Injury
MeSH Terms: conditions — Virus Diseases; Critical Illness; Multiple Organ Failure; Systemic Inflammatory Response Syndrome; Acute Kidney Injury | interventions — Hemoperfusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- EBP: ICU COVID-19 patients treated with hemoperfusion/hemadsorption
  Interventions: Device: Hemoperfusion
- non-EBP: ICU COVID-19 patients not treated with hemoperfusion/hemadsorption

INTERVENTIONS:
Device: Hemoperfusion — Commercial membranes for extracorporeal blood purification (hemoperfusion)
  Groups: EBP

SUMMARY:
The ongoing COVID-19 pandemic caused high hospitalization and mortality rates especially in critically ill patients. Unfortunately, there is no present study with a large number of patients that would offer us clear answers on the treatment of ICU COVID-19 patients with adsorption filters, extracorporeal methods and the hemoperfusion method. The purpose of this registry study is to investigate the effectiveness and safety of the extracorporeal blood purification and hemoperfusion/hemadsorption filters in treating of critically ill COVID-19 patients.

DETAILED DESCRIPTION:
The COVID-19 pandemic has been associated with high mortality rate and high percentage of patients with with severe multi-organ dysfunction. Many therapies were investigated in this group of patients. The usage of extracorporeal blood purification, namely hemoperfusion/hemadsorption was introduced in everyday clinical practice even before COVID-19 pandemic in which became increasingly common. The efficacy of hemoperfusion/hemadsorption in removal of endotoxins and cytokines is still questioned by some physicians mostly due to the fact that some trials failed to demonstrate the effect of this therapy on long-term outcomes of critically ill patients. Unfortunately, there is no present study with a large number of patients that would offer us clear answers on the treatment of ICU COVID-19 patients with adsorption filters, extracorporeal methods and the hemoperfusion method. Several extracorporeal blood purification therapies have been proposed to attenuate systemic inflammation in COVID-19 patients but there is no study which analyzed more than one filter or patients without specific conditions. Due to these limitations the studies were not able to analyze the method itself. Therefore, the primary aim of this observational prospective, multi-centric, regional web-based registry is to define the results and outcome of treatment, possible advantages over patients who have not undergone targeted treatment and to set regional indications/inclusion criteria for the treatment of ICU COVID-19 patients with the method of hemoadsorption/hemoperfusion.

ELIGIBILITY:
Inclusion Criteria:

1. COVID-19 infection
2. laboratory and clinical evidence of systemic inflammation: high levels of inflammatory cytokines such as IL-6 (>25 pg / ml); high values of inflammatory parameters from serum (leukocytes >15x10 9 / l, CRP >40 mg / l, procalcitonin >0.9 mg / l) and a high SOFA score (>2).
3. diagnosed with sepsis or septic shock: sepsis is defined as the presence of suspected or documented infections along with systemic inflammatory response syndrome; septic shock is defined as the presence of sepsis and acute circulatory failure according to European criteria Society for Intensive Care Medicine
4. clinical symptoms of hemodynamic instability requiring vasopressors and initial signs immune dysregulation or cascade coagulation disorders
5. acute kidney injury assessed according to KDIGO / AKIN criteria: increase in serum creatinine ≥ 0.3 mg / dL within 48 hours, or ≥ 50% over 7 days, or hourly diuresis <0.5 mL / kg / h for more than 6 hours
6. diagnosis of ARDS
7. the need for ECMO
8. deterioration of respiratory status with the onset of respiratory failure requiring mechanical ventilation (respiration rate >30 / min, or oxygen saturation <93%, or PaO2 / FiO2 ratio <300mmHg).
9. Admission to ICU

Exclusion Criteria:

* besides contraindications to the use of the hemoperfusion adopted (as from the manual of instructions), there are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All medical institutions from South-East European countries (Slovenia, Croatia, Bosnia, Montenegro, Serbia, Macedonia, Albania, Kosovo, Greece, Italy, Turkey, Bulgaria and Romania) that provide extracorporeal blood purification treatments to COVID-19 critically ill patients are eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Define the inclusion criteria for hemoperfusion in ICU COVID-19 patients | 28 days
  Define the inclusion criteria for extracorporeal blood purification (hemoperfusion) with different filters/hemadsorbers in ICU COVID-19 patients

SECONDARY OUTCOMES:
To assess the correlation between hemoperfusion and positive short-term outcome | 24 hours after hemoperfusion initiation
  Define as to assess the correlation between hemoperfusion and positive short-term outcome (i.e. an improvement in hemodynamic stability, inflammatory status and respiratory status).
To assess the correlation between hemoperfusion and positive short-term outcome | 72 hours after finishing all the hemoperfusion procedures
  Define as to assess the correlation between hemoperfusion and positive short-term outcome (i.e. an improvement in hemodynamic stability, inflammatory status and respiratory status).
To assess the correlation between hemoperfusion and positive long-term outcome | 28 days
  To assess the correlation between hemoperfusion and positive long-term outcome, defined as patient survival at ICU discharge.
To assess the correlation between different filters/hemadsorbers and positive short-term outcome | 24 hours after hemoperfusion initiation
  Define as to assess the correlation between different filters/hemadsorbers and positive short-term outcome (i.e. an improvement in hemodynamic stability, inflammatory status and respiratory status).
To assess the correlation between different filters/hemadsorbers and positive short-term outcome | 72 hours after finishing all the hemoperfusion procedures
  Define as to assess the correlation between different filters/hemadsorbers and positive long-term outcome (i.e. an improvement in hemodynamic stability, inflammatory status and respiratory status).
To assess the correlation between different filters/hemadsorbers and positive long-term outcome | 28 days
  To assess the correlation between different filters/hemadsorbers and positive long-term outcome, defined as patient survival at ICU discharge.
The effects of filters/hemadsorbents in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome | 24 hours after initiation of the procedure with the combination of filters/hemadsorbers and extracorporeal organ support therapy
  The effects of filters/hemadsorbents in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome (i.e. an improvement in hemodynamic stability, inflammatory status and respiratory status).
The effects of filters/hemadsorbents in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome | 72 hours after finishing all the procedures with the combination of filters/hemadsorbers and extracorporeal organ support therapy
  The effects of filters/hemadsorbents in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome (i.e. an improvement in hemodynamic stability, inflammatory status and respiratory status).
The effects of filters/hemadsorbents in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive long-term outcome | 28 days
  The effects of filters/hemadsorbents in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive long-term outcome (i.e. an improvement in hemodynamic stability, inflammatory status and respiratory status).

CONTACTS AND LOCATIONS:
Overall Officials: Vedran Premuzic, M.D., Ph.D., Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- University Hospital Center Zagreb, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lovric D, Situm I, Nedeljkovic V, Mogus M, Erceg A, Mazar M, Mihaljevic S, Premuzic V. Seraph(R) filter effectiveness in the treatment of circuit-related infections in ECMO patients-a single-center report. Front Med (Lausanne). 2025 Oct 17;12:1664552. doi: 10.3389/fmed.2025.1664552. eCollection 2025. PMID 41179859